CLINICAL TRIAL: NCT07031401
Title: Investigation of the Attitudes of Patients With Chronic Obstructive Pulmonary Disease Towards Traditional Complementary Medicine Practices
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: KutahyaHSU20250619
Record Dates: First submitted 2025-06-11; First posted 2025-06-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Nursing Care; Holistic Care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals with Chronic Obstructive Pulmonary Disease need the help and support of caregivers in issues such as limitations in their physical and social functions, inadequacy, social isolation, dependency, and continuing their daily lives. The World Health Organization (WHO) defines traditional medicine as knowledge, skills, and practices based on beliefs, experiences, and theories used for the prevention, diagnosis, recovery, and treatment of physical and mental disorders. Since traditional medicine varies from culture to culture, it covers different, unique treatments and practices of countries and even regions within countries. In some countries, these practices (CAM) are called 'alternative' and 'complementary'. There has been an increase in the use of complementary medicine in the last 30 years in developed and developing countries. While modern medical practices are used due to the supportive nature of complementary medicine, it is also used for purposes such as relaxing the patient, strengthening their immunity, and improving their psychological state. Patients diagnosed with COPD sometimes resort to alternative treatments. In parallel with the increase in life expectancy, the increase in chronic diseases such as COPD, which are difficult to care for and treat, the inability of healthcare professionals to allocate enough time, the suspicion of modern methods and possible side effects have greatly increased the interest in GETAT methods. The decrease in exercise capacity of COPD patients, frequent infection attacks, muscle weakness, and the accompanying anxiety and depression in these patients can be counted as reasons for increasing GETAT use. In light of this information, it was aimed to examine the attitudes of individuals with COPD towards GETAT use?

Research Questions; What is the GETAT use status of individuals with COPD? What are the attitudes of individuals with COPD towards GETAT?

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Must be 18 years or older
* Must be contactable

Exclusion Criteria:

*Those who are unable to communicate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Title: Determination of attitudes of individuals with COPD toward the use of Traditional and Complementary Medicine (TCM) | 6 months from the start of the study
  Description: Assessment of participants' attitudes toward Traditional and Complementary Medicine (GETAT in Turkish), using a validated attitude scale. The total attitude score will reflect the level of positivity or negativity in participants' perspectives.Time Frame: One-time assessment during data collectionAssessment Tool: Traditional and Complementary Medicine Attitude Scale (or equivalent validated tool in Turkish)Unit of Measure: Total attitude score (Likert scale)

SECONDARY OUTCOMES:
Frequency and type of TCM methods used by individuals with COPD | 6 months from the start of the study
  Description: Identification of which TCM methods (e.g., herbal medicine, acupuncture, cupping, etc.) are used, how frequently, and for what symptoms or purposes. One-time assessmentAssessment Tool: Researcher-developed questionnaire based on literatureUnit of Measure: Categorical data (Yes/No per method), frequency per month/year

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No